CLINICAL TRIAL: NCT06347861
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL, 3-PERIOD, 3-TREATMENT, 6-SEQUENCE, CROSSOVER, SINGLE-DOSE STUDY IN HEALTHY ADULT PARTICIPANTS TO ESTIMATE THE BIOAVAILABILITY OF THE REGISTRATION TABLETS OF VEPDEGESTRANT (ARV-471, PF-07850327) RELATIVE TO THE PHASE 3 TABLETS
Brief Title: A Study to Learn How Various Tablets of the Study Medicine Vepdegestrant Are Taken up Into the Blood of Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arvinas Estrogen Receptor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C4891003
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- single dose of vepdegestrant (3-period, 3-treatment, 6-sequence, crossover) (Experimental): Vepdegestrant administered as a single dose in Period 1, 2 and 3.
  Interventions: Drug: single dose of vepdegestrant as tablet formulation (Treatment A); Drug: single dose of vepdegestrant as tablet formulation (Treatment B); Drug: single dose of vepdegestrant as tablet formulation (Treatment C)

INTERVENTIONS:
Drug: single dose of vepdegestrant as tablet formulation (Treatment A) — phase 3 tablets
  Other Names: ARV-471, PF-07850327
Drug: single dose of vepdegestrant as tablet formulation (Treatment B) — registration tablets
  Other Names: ARV-471, PF-07850327
Drug: single dose of vepdegestrant as tablet formulation (Treatment C) — registration tablets
  Other Names: ARV-471, PF-07850327

SUMMARY:
The purpose of the study is to look at how various tablets of a study medicine called vepdegestrant are processed in the body. This will be studied in healthy adult participants after food.

This study looks at how the medicine is changed and removed from the body after a participant takes it.

This study is seeking for participant who:

* are healthy males, and healthy females who do not have the possibility to have children.
* are 18 years of age or older.
* weigh more than 45 Kilograms (99 pounds).

The study consists of 3 treatments. Each participant will be assigned by chance to receive the 3 treatments in a certain sequence. This will be done over 3 study periods. Each treatment consists of a single amount of vepdegestrant taken by mouth in each study period. There will be a washout period between each study periods. The washout period is the time allowed for the medicine to get washed out from the body. How the medicine was processed will be calculated following each dose in each period. The total study duration is about 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male participants and/or female participants of non-childbearing potential aged 18 years or older (or the minimum age of consent in accordance with local regulations) at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs and standard 12-lead ECGs.
* BMI of 16-32 kg/m2; and a total body weight >45 kg (99.2 lb).
* Capable of giving signed informed consent, which includes compliance with requirements and restrictions listed in the informed consent document (ICD) and in this protocol.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Participants with known history of sensitivity to vepdegestrant or any of the formulation components of vepdegestrant.
* Use of prescription or nonprescription drugs, including vitamins, dietary, herbal supplements, grapefruit/grapefruit containing products, and Seville orange/Seville orange containing products within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention. A longer washout is required for those that fall into the categories below:
* Moderate or strong CYP3A inducers which are prohibited within 14 days plus 5 half-lives prior to the first dose of study intervention.
* Moderate or strong CYP3A inhibitors which are prohibited within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention (unless otherwise indicated in the protocol).
* Standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) for vepdegestrant | Pre-dose, and 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, 120, 144, 168 hours post dose
Area under the curve from time zero to extrapolated infinite time [AUC (0 - ∞)] for vepdegestrant | Pre-dose, and 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, 120, 144, 168 hours post dose
  AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Time the participant provides informed consent through and including follow-up contact occurring 28 to 35 calendar days after the last administration of the study intervention.
Number of Participants With Clinical Laboratory Abnormalities | Time the participant provides informed consent through and including follow-up contact occurring 28 to 35 calendar days after the last administration of the study intervention.
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Time the participant provides informed consent through and including follow-up contact occurring 28 to 35 calendar days after the last administration of the study intervention.
Number of Participants With Electrocardiogram (ECG) Abnormalities | Time the participant provides informed consent through and including follow-up contact occurring 28 to 35 calendar days after the last administration of the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4891003